CLINICAL TRIAL: NCT03910049
Title: Does Indocyanine Imaging Scoring Predicts Postoperative PTH Levels at 24 Hours After Total Thyroidectomy
Brief Title: Does Indocyanine Imaging Scoring Predicts Postoperative Parathormone Levels at 24 Hours After Total Thyroidectomy
Acronym: ICGPREDICT
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Associate Professor in Surgery, Aristotle University Of Thessaloniki
Other Study IDs: ICG002
Record Dates: First submitted 2019-02-19; First posted 2019-04-10 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Thyroid; Parathyroid; Deficiency
Keywords: Indocyanine Green; Near Infrared Imaging; Total Thyroidectomy
MeSH Terms: conditions — Thyroid Diseases; Hypoparathyroidism | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: The group will include all adult patients that will sign ICF and will be operated for total thyroidectomy regardless of the undelying disease
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine green will be administered intravenously to patients enrolled in this study after the completion of total thyroidectomy in order to assess the visibility of parathyroid glands and to assess the possible correlation of ICG score with post-operative parathormone levels in order to predict post-thyroidectomy hypoparathyroidism.
  Other Names: indocyanine green solution

SUMMARY:
The aim of the present study is to evaluate the prognostic value of intra-operative indocyanine staining scoring concerning 24 hours post-operative PTH levels and the possible advantages that its' use can give in terms of clinical practice compared to conventionally operated patients.

DETAILED DESCRIPTION:
Study objectives are:

* Detecting the changes of practice in performing total thyroidectomy with ICG.
* Comparing ICG-performed minimal invasive total thyroidectomy
* Identifying the cut-off points that predict low PTH levels (less than 20pg/ml)
* Identifying and analyzing problematic groups of patients The study is designed as a prospective observational multi-center study. Any patient that has indication for a total thyroidectomy will be considered eligible.

The study will be conducted until 60 subjects are included. It is estimated that it will take up to 3 months to enroll the patients.

Pre-Surgery: Procedures preformed such as routine hospital examinations, antibiotic prophylactic treatment, anticoagulant treatment and diet will be according to the standard management protocol and will be recorded for the study. The following pre-surgery information will be recorded:

1. Demographic information including: name, age, gender, ethnicity
2. Height, weight, BMI and American Society of Anesthesiologists physical status classification system (I-VI)
3. Behavioral history (Smoking, alcohol or drug use)
4. Preoperative labs (WBC, Ht, Hgb, Ca2+, P, fT3, fT4, TSH, PTH, VitD)
5. Diagnosis including clinical observations and previous imaging results
6. Pre-operative characteristics of the adenoma
7. Medications
8. Current and past history of surgical and medical comorbidities

Intra-operative: The surgeon will perform the preplanned operation. The following intraoperative variables will be recorded for all patients:

1. Surgery date
2. Duration of surgery
3. Operation performed
4. Procedure related comments
5. Number and location of the visualized glands
6. Intra-operative ICG score (ranging from 1 to 3 [5]) for each grand

Pathology data form: The following pathology data will be recorded for all patients:

1. Post-operative diagnosis including pathology report
2. Possible parathyroids excised Postoperative follow-up: Follow-up evaluation will be performed during hospitalization

1 Postoperative labs (WBC, Ht, Hgb, Ca2+, P, fT3, fT4, TSH, PTH)

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years old
* Patient scheduled for a non-emergency operation
* Patient eligible for total thyroidectomy

Exclusion Criteria:

* Patient is participating in another clinical trial which may affect this study's outcomes
* Prior operation in the neck
* Primary or secondary hyperparathyroidism
* Vitamin D deficiency
* Use of drugs that influences calcium metabolism (Vitamin D analogues, oral calcium supplements, bisphosphonates, teriparatide, thiazide diuretics, aromatase inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are going to have a total thyroidectomy regardless of the underlying pathology
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Intra-operative ICG fluarangiography predicts post-operative PTH values | 24 hours
  Whether ICG score of parathyroid glands after total thyroidectomy correlates with 24 post-operative values of PTH

SECONDARY OUTCOMES:
ICG improves the intraoperative recognizability of the parathyroids | Intraoperative
  To assess the ability of ICG flurangiography to increase recognizability of parathyroid glands during total thyroidectomy based on ICG score of the parathyroids.

CONTACTS AND LOCATIONS:
Overall Officials: Theodosios S Papavramidis, PhD, Study Director — Assistant Professor of Surgery
Locations (2):
- Greece (2):
  - Unit of Endocrine Surgery, Interbalkan Medical Center, Thessaloniki, Greece, Thessaloniki, Please Enter the State Or Province
  - 1st Propedeutic Department of Surgery, AHEPA University General Hospital, Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided